CLINICAL TRIAL: NCT07030478
Title: A Phase I/IIa Study to Evaluate the Safety and Tolerability of Monoclonal Antibody EP0089 in Patients With Advanced Solid Tumours
Brief Title: A Study to Evaluate the Safety and Tolerability of EP0089
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ellipses Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0089-101
Record Dates: First submitted 2025-05-30; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Solid Cancers; Solid Tumours

STUDY DESIGN:
Intervention Model Description: The trial is open-label with dose-escalation, and dose optimisation/expansion components to evaluate the safety, tolerability, and preliminary anti-tumour activity of EP0089.
  The starting dose and schedule for the planned dose escalations have been carefully selected based on preclinical data, and in line with relevant regulatory standards, using a standard 3+3 dose escalation design for all dose levels with the exception of dose level 1 which will apply to a single patient only. Specific safety evaluations are included to evaluate potential toxicities identified in preclinical toxicity studies. The study also includes a thorough assessment of PK/PD and evaluation of the impact of biomarkers to evaluate potential patient selection strategies and establish proof of mechanism.
Masking Description: N/A - is an open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): 3+3 design evaluating the safety and efficacy of EP0089
  Interventions: Drug: EP0089-101

INTERVENTIONS:
Drug: EP0089-101 — EP0089 will be initially administered by intravenous (IV) infusion once every 2 weeks (Q2W)

SUMMARY:
This is a first-in-human (FIH), first-in-class, Phase I/IIa, open-label study designed to evaluate the safety and tolerability of EP0089 (study drug). Study drug will initially be given via intravenous (IV) infusion once every 2 weeks (Q2W), with one treatment cycle defined as 14 days. The study will enroll patients with advanced solid tumours for whom no standard therapy exists or for whom standard therapy has failed. An independent Safety Monitoring Committee (SMC) will review safety data at regular intervals to ensure participant safety and support dose escalation decisions.

ELIGIBILITY:
Inclusion Criteria:

Applicable to all patients:

1. Must be ≥18 years of age (≥19 in South Korea) with documented recurrent, metastatic or unresectable solid tumours for whom no standard therapy exists or standard therapy has failed
2. ECOG performance status of 0 or 1 and life expectancy >3 months at screening
3. Ability to understand and provide written informed consent
4. Must be willing to comply with necessary contraceptive methods as required
5. Willing and able to comply with the scheduled study treatment plan, laboratory tests, and other study procedures.
6. Adequate hepatic, haematological and renal function as assessed by protocol-defined criteria.
7. Additional cohort/disease specific criteria apply
8. Measurable disease per RECIST v1.1

Exclusion Criteria:

1. Known active CNS metastases and/or leptomeningeal disease and/or carcinomatous meningitis.
2. Recent major surgery
3. Recent live or live-attenuated vaccine ≤ 30 days prior to the first dose
4. Current active, or history of, autoimmune disease that requires or required systemic treatment (ie, with disease modifying agents, corticosteroids, or immunosuppressive drugs) within 2 years prior to starting study treatment.
5. Prior severe hypersensitivity reaction to mAbs
6. Previous > Grade 2 peripheral neuropathy.
7. Significant neurological condition eg stroke, transient ischaemic attack (in the last 12 months), epilepsy, head trauma, brain surgery or prior history of any significant psychiatric disorder

9. Current active, or history of, autoimmune disease that requires or required continuous treatment within 2 years prior to starting study treatment

10. Receiving chronic systemic steroid therapy (> 10 mg /day of prednisone or equivalent) or any other form of immunosuppressive therapy ≤ 7 days prior the first dose of study drug. Topical or inhaled steroids are permitted.

11. Any prior immune-mediated or immune-related adverse events related to treatment with immune-modulatory agents that caused permanent discontinuation of the agent, that were ≥ Grade 3 in severity or in the opinion of the Investigator would otherwise jeopardise patient safety in this study.

12. One or more clinically significant (ie, active) cardiovascular diseases, myocardial infarction, or unstable angina (≤ 6 months prior to first administration of study drug)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of EP0089 | 126 weeks
  The study's main goal is to find the highest safe dose of EP0089 and the best dose for future testing.

IPD SHARING:
Plan to Share IPD: No